CLINICAL TRIAL: NCT05516888
Title: A Prospective, Randomized Comparison of the Radiofrequency of Gasserian Ganglion Versus Peripheral Branches of the Trigeminal Nerve for the Treatment of Trigeminal Neuralgia.
Brief Title: Comparison of the Radiofrequency Treatments for the Treatment of Trigeminal Neuralgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 138/14
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency of peripheral branches of the trigeminal nerve (Experimental): pulsed radiofrequency treatment of the peripheral branches of the trigeminal nerve
  Interventions: Procedure: radiofrequency of the peripheral trigeminal branches
- Radiofrequency of gasserian ganglion (Active Comparator): radiofrequency ablation of the gasserian ganglion
  Interventions: Procedure: radiofrequency of gasserian ganglion

INTERVENTIONS:
Procedure: radiofrequency of gasserian ganglion — radiofrequency ablation of the gasserian ganglion
  Arms: Radiofrequency of gasserian ganglion
Procedure: radiofrequency of the peripheral trigeminal branches — radiofrequency of the peripheral trigeminal branches ( maxillary, mandibular, supraorbital)
  Arms: Radiofrequency of peripheral branches of the trigeminal nerve

SUMMARY:
The aim of this study is to compare the efficacy of radiofrequency of the Gasserian ganglion versus peripheral branches of the trigeminal nerve for the treatment of trigeminal neuralgia.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is defined as sudden, severe, short-term, stabbing and recurrent pain in the distribution of one or more branches of the trigeminal nerve. Many invasive treatments are available for patients who respond poorly to medical therapy. Among them, radiofrequency therapy is a viable option with a reliable initial and long-term clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Primary Trigeminal Neuralgia meets the criteria of the International Classification of Headache Disorders.
* Suffering from severe trigeminal neuralgia that cannot be alleviated effectively with conservative therapy.
* Agree to participate in the study

Exclusion Criteria:

* Infection at the puncture site.
* Coagulation disorder.
* Abnormal blood test (hepatic or renal function)
* History of receiving invasive treatment (glycerol rhizolysis, radiofrequency thermocoagulation, balloon compression, gamma knife treatment, microvascular decompression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
The modified Barrow Neurological Institute Pain Intensity Score | six months
  The efficacy of the treatment will be assessed using the modified Barrow Neurological Institute Pain Intensity Score (I: No pain, off medications; II: Occasional pain, off medications; IIIa: No pain, continued use of medications; IIIb: Pain persists, but adequately controlled with medications; IV: Pain not adequately controlled with medications; V: No relief).

SECONDARY OUTCOMES:
Numeric rating scale | baseline to six months
  Pain will evaluated by a numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable).
Patient satisfaction | six months
  Patient satisfaction scores on the 5-point Likert scale (1: poor, 2: fair, 3: good, 4: very good, 5: excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)